CLINICAL TRIAL: NCT06349486
Title: Efficacies of Bismuth-amoxicillin-vonoprazan Triple Therapy, Vonoprazan-amoxicillin Dual Therapy and Proton Pump Inhibitor-based Standard Triple Therapy in the First-line Anti-H. Pylori Treatment
Brief Title: Efficacies of Bismuth-amoxicillin-vonoprazan Triple Therapy, Vonoprazan-amoxicillin Dual Therapy and Proton Pump Inhibitor-based Standard Triple Therapy for Hp Eradication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, DENG-CHYANG WU, clinical professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20230179
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-04

CONDITIONS: Helicobacter Pylori Eradication
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Rabeprazole; Clarithromycin

STUDY DESIGN:
Intervention Model Description: 1. bismuth-amoxicillin-vonoprazan triple therapy
  2. vonoprazan-amoxicillin dual therapy
  3. proton pump inhibitor-based standard triple therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bismuth-amoxicillin-vonoprazan triple therapy (Active Comparator): vonoprazan 20mg twice a day + amoxicillin 750mg four times a day + tripotassium dicitrate bismuthate 300mg four times a day
  Interventions: Drug: vonoprazan, amoxicillin, tripotassium dicitrate bismuthate
- vonoprazan-amoxicillin dual therapy (Active Comparator): vonoprazan 20mg twice a day + amoxicillin 750mg，Four times a day
  Interventions: Drug: vonoprazan, amoxicillin
- proton pump inhibitor-based standard triple therapy (Active Comparator): rabeprazole 20mg twice a day + amoxicillin 1gm twice a day + clarithromycin 500mg twice a day
  Interventions: Drug: rabeprazole, amoxicillin, clarithromycin

INTERVENTIONS:
Drug: vonoprazan, amoxicillin, tripotassium dicitrate bismuthate — bismuth-amoxicillin-vonoprazan triple therapy
  Arms: bismuth-amoxicillin-vonoprazan triple therapy
Drug: vonoprazan, amoxicillin — vonoprazan-amoxicillin dual therapy
  Arms: vonoprazan-amoxicillin dual therapy
Drug: rabeprazole, amoxicillin, clarithromycin — proton pump inhibitor-based standard triple therapy
  Arms: proton pump inhibitor-based standard triple therapy

SUMMARY:
1. Compare the efficacies and safety of 14-day bismuth-amoxicillin-vonoprazan tiple therapy, 14-day vonoprazan dual therapy and 14-day rabeprazole triple therapy in the first-line treatment of H. pylori infection.
2. To investigate the impacts of antibiotic resistance of H. pylori as well as CYP3A4, CYP2C19 and IL-1B -511 genotypes of host on the eradication efficacies of anti-H. pylori treatments.

DETAILED DESCRIPTION:
For this multi-center, randomized, open-label, superiority trial, we will recruit 780 adult patients with H. pylori infection from ten medical centers or regional hospitals in Taiwan. Using a computer generated randomized sequence, we randomly allocate patients (1:1:1; block size of six) to either 14-day bismuth-amoxicillin-vonoprazan triple therapy, 14-day vonoprazan dual therapy, or 14-day rabeprazole-triple therapy. Patients are asked to return at the second week to assess drug adherence and adverse events. Post-treatment H. pylori status is assessed by 13C-urea breath test at week 6. Participants with failure of H. pylori eradication will randomly receive either 14-day vonoprazan-based or 14-day esomeprazole-based bismuth quadruple therapy. Finally, the rates of eradication and adverse events will be compared between groups by chi-square test. Additionally, the effects of antibiotic resistances of H. pylori as well as CYP3A4, CYP2C19 and IL-1B -511 genotypes of host on the eradication efficacies of above first-line and second-line anti-H. pylori treatments are assessed by multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

(1) At least 18 years old. (2) Subjects infected with Helicobacter pylori.

Exclusion Criteria:

1. Those who have ever received Helicobacter pylori sterilization treatment.
2. Those who are allergic to the drugs used in this research.
3. Those who have had stomach surgery.
4. Those with severe liver cirrhosis or uremia or malignant tumors.
5. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the eradication rate of Helicobacter pylori | 8 week after finishing study drugs
  evalute eradication outcome by 13C urea breath test

SECONDARY OUTCOMES:
genotype analysis | 1 day
  CYP3A4, CYP2C19 and IL-1B -511 genotypes

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan